CLINICAL TRIAL: NCT02173080
Title: Development and Assessment of the Psychometric Properties of a Polycystic Liver Disease-specific Patient Reported Outcomes Questionnaire (PLD-Q).
Brief Title: Development and Assessment of The Polycystic Liver Disease Questionnaire (PLD-Q).
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marie Hogan, PI, Mayo Clinic
Other Study IDs: 14-003832
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Polycystic Liver Disease
Keywords: autosomal dominant polycystic liver disease; autosomal dominant polycystic kidney disease; quality of life; patient reported outcome tool
MeSH Terms: conditions — Polycystic liver disease; Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Polycystic liver disease patients: will receive PLD-Q, EORTC QLQ-30 symptoms subscale, EQ5D-VAS score and SF36
  Interventions: Other: PLD-Q
- ADPKD group without PLD: will receive PLD-Q
- Healthy controls: receive PLD-Q
  Interventions: Other: PLD-Q
- PLD patient focus group: to discuss and improve PLD-Q
- PLD clinical expert focus group: to discuss and improve PLD-Q

INTERVENTIONS:
Other: PLD-Q — polycystic liver disease questionnaire
  Groups: Healthy controls; Polycystic liver disease patients

SUMMARY:
This Pilot study will enable development & assessment of a Polycystic Liver Disease-specific patient reported outcomes questionnaire (PLD-Q). Polycystic liver disease (PLD) is characterized by the formation of numerous cysts in the liver, and can lead to severe symptomatic hepatomegaly. It is common in patients with autosomal dominant polycystic liver disease (ADPLD) and autosomal dominant polycystic kidney disease (ADPKD).

DETAILED DESCRIPTION:
As liver function is preserved, quality of life is the main outcome in PLD. Patient reported outcomes are increasingly utilized to assess treatment efficacy & can include any endpoint derived from patient reports & are usually assessed by questionnaire. Several existing generic questionnaires assess gastrointestinal symptoms, but include irrelevant items for polycystic liver disease (PLD) & do not examine relevant extra-abdominal symptoms. Also, a questionnaire that assesses the full range of PLD related problems is more likely to be responsive to changes after treatment initiation. Therefore, a tool that accurately detects changes in PLD symptoms is required.

The development and first steps of validation of this questionnaire are already completed in Netherlands. We will further develop this questionnaire for English speaking patients and validate it in Mayo Clinic cohorts.

The study contains three phases. Phase 1: pilot testing of the directly translated questionnaire (from dutch into english) in a small group of polycystic liver disease (PLD) patients. We will include both symptomatic & asymptomatic patients (i.e. from mild to severe PLD). Phase 2: further refinement of the questionnaire using the results of the pilot test and input of Mayo patient and clinician focus groups. Phase 3: Further validation in a large cohort of 200 PLD patients with (1) comparison with 200 controls without PLD, (2) cross-sectional correlation with total liver (TLV) & kidney volumes (TKV), (3) comparing ADPKD patients with & without PLD (5) against other validated questionnaires (e.g. SF36) & (5) development of a custom "Worry Questionnaire" examining disease-related worries & concerns. Finally, longitudinal analyses will be performed to assess PLD-Q sensitivity to change in symptoms. Statistical & psychometric analyses will be provided by Mayo Clinic quality of life Research group, & developed in accordance with Food and Drug Administration (FDA) guidance on patient-reported outcome measures in consultation with their Study Endpoints & Labeling Development Division.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 year
* Polycystic liver, defined by > 20 liver cysts on imaging

Exclusion Criteria:

* Patients unable to speak or read the English properly
* History of kidney or liver transplantation
* Dialysis
* Current use of experimental drugs (e.g. lanreotide, octreotide)
* Recent liver resection or major surgery
* Other comorbidities that can affect the outcome of the questionnaire, as deemed by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with polycystic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 594 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Polycystic Liver Disease-specific patient reported outcomes questionnaire (PLD-Q) total score | baseline to 6 months
  total score on the PLD-Q

SECONDARY OUTCOMES:
The Short Form (36) Health Survey (SF36) | baseline to 6 months
European Organisation for Research and Treatment of Cancer Quality of life questionnaire (EORTC-QLQ-C30) symptom subscale | baseline to 6 months
Euroqol group 5 dimensions questionnaire visual analog score (EQ5D-VAS) | baseline to 6 months
Total liver volume | baseline
Total kidney volume | baseline
  measured in patients with autosomal dominant polycystic kidney disease (ADPKD)

CONTACTS AND LOCATIONS:
Overall Officials: Marie C Hogan, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials